CLINICAL TRIAL: NCT04951492
Title: Olaparib in Prostate Cancer Patients With Evidence of Homologous Recombination Deficiency as Assessed Using an Integrated Genomic Signature
Brief Title: Olaparib for the Treatment of Castration Resistant Prostate Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawal of funding
Sponsor: University of Washington (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Michael Schweizer, Associate Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1121519; NCI-2021-06147 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RG1121519 (Other: Fred Hutch/University of Washington Cancer Consortium); 10759 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2021-06-28; First posted 2021-07-06 (Actual); Results first posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Castration-Resistant Prostate Carcinoma; Prostate Adenocarcinoma
MeSH Terms: interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Olaparib) (Experimental): Patients receive olaparib orally (PO) twice daily (BID). Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU-0059436; Lynparza; PARP Inhibitor AZD2281

SUMMARY:
This phase II trial investigates the effect of olaparib in treating patients with castration resistant prostate adenocarcinoma. Olaparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive olaparib orally (PO) twice daily (BID). Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol
* Subject must be >= 18 years of age at the time of signing the informed consent form
* Individuals who have documented histologically confirmed adenocarcinoma of the prostate
* Subject must have evidence of castration resistant prostate cancer as evidenced by PSA progression (per Prostate Cancer Working Group 3 [PCWG3] criteria) and a castrate serum testosterone level (i.e. =< 50 mg/dL)
* PSA must be at least 2 ng/mL and rising on two successive measurements at least two weeks apart
* At least one lesion (measurable and/or non-measurable) that can be accurately assessed at baseline by computed tomography (CT) scan, magnetic resonance imaging (MRI), or positron emission tomography (PET) and is suitable for repeated assessment
* Must have progressed on abiraterone and/or a second-generation androgen receptor (AR) antagonist (i.e. enzalutamide, apalutamide, or darolutamide). If these were given in the hormone sensitive setting, patients must also have progressed on at least one prior approved therapy for CRPC
* Must have archival tissue available or be willing to undergo metastatic biopsy in order to perform next-generation deoxyribonucleic acid (DNA) sequencing and undergo whole exome sequencing
* Patient must have a positive LOH score on prior University of Washington (UW) OncoPlex testing
* Hemoglobin >= 10.0 g/dL with no blood transfusion in the past 28 days (within 28 days prior to administration of study treatment)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (within 28 days prior to administration of study treatment)
* Platelet count >= 100 x 10^9/L (within 28 days prior to administration of study treatment)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (within 28 days prior to administration of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be =< 5 x ULN (within 28 days prior to administration of study treatment)
* Patients must have creatinine clearance estimated of >= 51 mL/min using the Cockcroft-Gault equation or based on a 24 hour urine test (within 28 days prior to administration of study treatment)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patients must have an estimated life expectancy >= 16 weeks
* Male patients must use a condom during treatment and for 3 months after the last dose of olaparib when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential

Exclusion Criteria:

* As judged by the investigator, any evidence of serious and/or unstable pre-existing medical or psychiatric condition which in the investigator's opinion makes it undesirable for the patient to participate in the trial
* Other malignancy unless curatively treated with no evidence of disease for >= 5 years except: adequately treated non-melanoma skin cancer and non-muscle invasive bladder cancer
* Resting electrocardiography (ECG) indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, corrected QT interval by Fridericia's formula [QTcF] prolongation > 500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome
* Persistent toxicities (> Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia
* Patients with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML)
* Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on high resolution computed tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV) and are not receiving active treatment or have a detectable viral load
* Patients with known active hepatitis (i.e. hepatitis B or C).

  * Active hepatitis B virus (HBV) is defined by a known positive HBV surface antigen (HBsAg) result. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody and absence of HBsAg) are eligible
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA)
* Any previous treatment with PARP inhibitor, including olaparib
* Any previous treatment with platinum chemotherapy in the metastatic castration-resistant setting
* Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment
* Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks
* Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's wort ) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product
* Involvement in the planning and/or conduct of the study
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schweizer, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Olaparib)
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Olaparib)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Lowest On-treatment Prostate Specific Antigen (PSA)
Description: The proportion of patients achieving at least a 50% decline in PSA from baseline will be presented.
Time Frame: At least 12 weeks of olaparib treatment
Population: Patients who received at least 12 weeks of olaparib
Measure: Number; unit: participants
Arm/Group | Treatment (Olaparib)
Number analyzed (Participants) | 1
participants | 0

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Will be defined as the proportion of participants demonstrating at least a 30% decrease in total tumor size from baseline per Response Evaluation Criteria in Solid Tumors 1.1 criteria at any time point. The percent of patients with ORR and range of values will be provided.
Time Frame: Up to 12.3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Olaparib)
Number analyzed (Participants) | 2
Participants | 0

3. Secondary Outcome: Radiographic Progression Free Survival (PFS)
Description: Radiographic progression will be determined as using RECIST v1.1 and/or PCWG3 criteria. Median PFS will be estimated using the Kaplan-Meier method.
Time Frame: Up to 12.3 weeks
Measure: Median (Full Range); unit: weeks
Arm/Group | Treatment (Olaparib)
Number analyzed (Participants) | 2
weeks | 12.3 [11 to 12.3]

4. Secondary Outcome: Prostate Specific Antigen (PSA) Progression Free Survival (PFS)
Description: PSA progression will be time to for the PSA to increase by at least 2 ng/ml and ≥20% above baseline. PSA PFS will be the time until PSA progression and will be analyzed using kaplan meier method, with the median PSA PFS reported
Time Frame: Up to 16.6 weeks
Measure: Median (Full Range); unit: weeks
Arm/Group | Treatment (Olaparib)
Number analyzed (Participants) | 2
weeks | 12 [12 to 16.6]

5. Secondary Outcome: Overall Survival
Description: Number of patients who died on study. Note: Plan was to assess time from enrollment to death; however, no deaths have been observed.
Time Frame: Up to 12.3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Olaparib)
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: Within 30 days of end of treatment, up to 16.6 weeks
Arm/Group | Treatment (Olaparib)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Olaparib) (N=2)
Pulmonary Embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Olaparib) (N=2)
Nausea (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Left Forearm Tear (Injury, poisoning and procedural complications) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Lightheadedness (Nervous system disorders) | 1 (1)
White Blood Cell Count Decreased (Investigations) | 1 (1)
Neutrophil Count Decreased (Investigations) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT04951492/Prot_SAP_002.pdf
  • Informed Consent Form (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT04951492/ICF_000.pdf